CLINICAL TRIAL: NCT00604253
Title: Comparison of Efficacy and the Safety of Insulin Detemir and Insulin NPH as add-on to Current OHA Therapy in Subjects With type2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Insulin Detemir in Type 2 Diabetes Inadequately Controlled on OHA Therapy Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1477; JapicCTI-R070009 (Registry Identifier: japic)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the efficacy of insulin detemir on blood glucose control in type 2 diabetes when added to current OHA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Duration of type 2 diabetes mellitus for at least one year
* Insulin naive patients
* OHA treatment for at least 12 weeks
* HbA1C between 7.5-10.0%
* Body Mass Index (BMI) below 30.0 kg/m2

Exclusion Criteria:

* Impaired renal function
* Impaired hepatic function
* Pregnant, breast-feeding (within a year after delivery), intention of becoming pregnant or not using adequate contraceptive methods

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2003-12; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 36 weeks of treatment

SECONDARY OUTCOMES:
Plasma glucose profiles
Incidence of hypoglycaemic episodes
Adverse events
Insulin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Kobayashi M, Iwamoto Y, Kaku K, Kawamori R, Tajima N. 36-week Randomized Multicenter Open-label Parallel Group Phase 3 Trial to Compare Insulin Detemir and NPH Insulin Efficacy and Safety in Once Daily Treatment as an Add-on Current Oral Hypoglycemic Agents. J. Japan Diab. Soc 2007; 50 (9): 665-677
- [Result] Tajima N, Iwamoto Y, Kaku K, Kawamori R, Nishida T, Kobayashi M. Once-daily insulin detemir added to oral antidiabetic drugs results in less weight gain and a trend for reduced hypoglycaemia in comparison with NPH insulin in Japanese patients with type 2 diabetes. Diabetologia 2006; 49 (Suppl. 1): 609 (Abstract 996)
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com